CLINICAL TRIAL: NCT04726449
Title: Observatory of Psychiatric Symptoms and Their Somatic Causes in Urgent Medical Care (OPOSSUM)
Brief Title: Observatory of Psychiatric Symptoms and Their Somatic Causes in Urgent Medical Care
Acronym: OPOSSUM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1071
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-07

CONDITIONS: Neurologic Disorder; Psychiatric Disorder
MeSH Terms: conditions — Nervous System Diseases; Mental Disorders | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psychiatric diagnosis: psychiatric diagnosis : patients who were given a psychiatric diagnosis at the end of the follow up
  Interventions: Other: Screening for acute confusional state
- somatic diagnosis: somatic diagnosis: patients who were given a somatic diagnosis at the end of the follow up
  Interventions: Other: Screening for acute confusional state

INTERVENTIONS:
Other: Screening for acute confusional state — The intervention will consist of two psychometric test to screen for acute confusional state with the usual physical examination by the emergency physician. The neurological examination abnormalities will be noted

SUMMARY:
Use of emergency department for psychiatric symptoms always addresses the question of a potential somatic cause to the symptoms. Despite the wide-spread use of standard biology test and systematic brain imaging (for a first episode), there are still up to 5% of patients sent in psychiatric wards that actually have a somatic explanation to their symptoms which induces an important delay in the diagnostic assessement We hypothesized that simple neurological clinical examination along with fast psychometric screening tests in the Emergency Room (ER) could help the physicians to better screen the patients and thus prevent inaccurate post-emergency orientation.

Every patient visiting the ER for psychiatric symptoms will be included. The usual physical examination by the ER physician will be associated with two psychometric tests (namely the Clock-drawing test and Frontal Assessment Battery test).

The follow up will be made after 3 months in order to have the final diagnosis. Neurological data and data from the FAB test and the Clock-drawing test will be compared between patients who were finally given a psychiatric diagnosis versus patients with a somatic diagnosis at the end of the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Patient consulting the emergency room for psychiatric recourse
* Benefiting from a consultation with a psychiatrist in the emergency room
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient objecting to the conduct of this study and the collection of health data
* Patient with motor disorders preventing the performance of a test requiring a pencil
* Patient sedated before treatment in the emergency room
* Patient with visual disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient using emergency department for a psychiatric symptom
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Somatic or psychiatric nature of the final diagnosis given to the patient | At 3 month
  interview patient to collect during the last 90 days the data of a hospitalization, its possible duration, the examinations that may have been necessary to obtain the diagnosis: blood, urine, Cerebrospinal Fluid, imaging exams, electroencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: KARIM TAZAROURTE, MD, PhD, Principal Investigator — Hôpital Edouard Herriot, HCL
Locations (1):
- Service Accueil des Urgences, Hopital Edouard Herriot, Lyon, Rhône, France